CLINICAL TRIAL: NCT07275931
Title: Digital Support Program Via 1177 for Patients With Heart Failure - a Cluster-Randomized Hybrid Type 2 Study for Evaluation of Effects and Implementation
Brief Title: Digital Support Program for Patients With Heart Failure - a Cluster-Randomized Hybrid Type 2 Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Anna Stroemberg, Professor, Linkoeping University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023-04289-01
Record Dates: First submitted 2025-11-26; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Heart Failure With Reduced Ejection Fraction
Keywords: Co-design; E-health; support; implementation; RE-AIM; PRISM; ERIC

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tailored implementation (Experimental): This arm will receive tailored implementation support.
  Interventions: Other: Tailored implementation support
- Control (No Intervention): This group will receive standard implementation of the support program.

INTERVENTIONS:
Other: Tailored implementation support — Tailored implementation support
  Arms: Tailored implementation

SUMMARY:
The overall aim of this project is to evaluate the effects of a digital support program for patients with heart failure through a cluster-randomized controlled trial, and to investigate the outcomes of different implementation strategies using the RE-AIM (Reach, Effectiveness, Adoption, Implementation, Maintenance), PRISM (Practical, Robust Implementation and Sustainability Model) and ERIC (Expert Recommendations for Implementing Change) framework.

Our primary hypothesis is that the digital support program will improve patients' perceived control over their heart failure, measured with the validated Control Attitude Scale.

Secondary hypotheses are that the program will increase patients' health-related quality of life, self-care behaviors, heart failure knowledge, perceived continuity of care, and participation in care, and reduce symptoms of depression.

Implementation aim (based on the RE-AIM, PRISM and ERIC frameworks) The implementation component of the study aims to compare two different implementation strategies: a standard (basic) support package versus a tailored, context-specific support strategy.

Heart failure clinics at hospitals an within primary care will be matched and randomized into two arms. The intervention arm will receive tailored implementation support to implement the support program. The control arm will recive implementation support according to a predefined standard procedure.

Researchers will compare the intervention arm with control arm to see if there are any differences regarding the implementationsuccess between the arms.

The patients in both arms will have access to the support program during six months.

DETAILED DESCRIPTION:
Will be added

ELIGIBILITY:
Inclusion criteria:

* Diagnosed with heart failure with reduced ejection fraction (HFrEF) or heart failure with midrange reduced ejection fraction (HFmrEF) (ejection fraction ≤50%) verified by echocardiography or Magnetic Resonance Imaging
* Access to BankID, a computer, tablet, or smartphone
* Aged ≥18 years
* Able to understand and communicate in Swedish
* Provided informed consent

Exclusion criteria:

* Barriers to participation (e.g., not Swedish-speaking, cognitive impairment, severe mental illness, substance abuse)
* Life expectancy of less than six months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Perceived control attitudes | At enrollment and at the end of the intervention at 6 month
  Measured with The Control Attitudes Scale-Revised. The scale has 8 item. The possible range for the total score is from 8 to 40. Higher scores reflect greater levels of perceived control.

SECONDARY OUTCOMES:
Self-care | At enrollment and at the end of the intervention at 6 month
  Measured using the European Heart Failure Self-care Behaviour Scale. The scale has 9 item. The possible range for the total score is from 0 to 100. Higher scores reflect greater levels of self-care.
Perceived control | At enrollment and at the end of the intervention at 6 month
  Perceived Attitude Scale with 4 items. The possible range for the total score is from 4 to 28. Higher scores reflect higher levels of perceived control.
Heart failure knowledge | At enrollment and at the end of the intervention at 6 month
  Heart failure knowledge scale has 3 parts. The first part has 15 knowledge questions and the possible range for the total is 0-15. Higher scores reflect greater levels of knowledge. The second part measures the trust the person with heart failure has in his/her knowledge with 3 items on a scale from 1-5 and the possible range for the total is 3-15. Higher scores reflect greater levels of trust.The third part measures perception of knowledge with 3 items on a scale from 1-5 and the possible range for the total is 3-15. Higher scores reflect greater levels of perceived knowledge.
Healthcare consumtion | From enrollment to 12 month follow-up
  Patient records of all health care consumption
Health related quality of life | At enrollment and at the end of the intervention at 6 month
  Measured with Euro-Qol EQ-5D, The scale has 6 item. The first 5 items comprises 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The digits for the 5 dimensions can be combined into a 5-digit number that describes the patient's health state.
  Item 6 is a Visual Analog Scale. The possible range for the total score is from 0 to 100. Higher scores reflect greater levels of health.
Disease specific health-related quality of life | At enrollment and at the end of the intervention at 6 month
  Measured with Kansas City Cardiomyopathy questionnaire. The scale has 12 items assessing 4 domains (physical limitation, symptom frequency, quality of life, and social limitation), which can be reported separately into the subscales or summed into an overall score. The scales range from 0 to 100, with higher scores indicating a better health status and low symptom burden.
Symptoms of Depression | At enrollment and at the end of the intervention at 6 month
  Measured with Patient Health Questionnare 9. The questionnaire has 9 items. The possible range for the total score is from 0 to 27. Higher score indicate more severe symptoms of depression.
Continuity of care | At enrollment and at the end of the intervention at 6 month
  Measured with Patient experiences continuity of care with 20 items on continuity of care in 4 dimensions: information, relations, management and knowlegde. The possible range for the total score is from 20 to 80. Higher score indicate better continuity.
Electronic Health Literacy | At enrollment and at the end of the intervention at 6 month
  Measured with Electronic health literacy scale. This scale contains 8 items and covers 3 dimensions: the ability to acquire, evaluate, and apply health information online. The scale uses a 5-point Likert scale, with responses ranging from 1 ("strongly disagree") to 5 ("strongly agree"). The total score ranges from 8 to 40, with higher scores indicating higher levels of electronic health literacy.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Stroemberg, Principal Investigator — Linkoeping University
Locations (1):
- Linköping University Hospital, Linköping, Östergötland County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Link to the support program — https://liu.se/forskning/digitalt-stodprogram-leva-med-hjartsvikt